CLINICAL TRIAL: NCT03904628
Title: Single-center, Dose Escalation, Open Phase I Clinical Study of Oral TG02 Capsule in the Treatment of Recurrent / Progressive High-grade Glioma Patients With Failed TMZ Treatment
Brief Title: Phase I Clinical Study of Oral TG02 Capsule in the Treatment of Recurrent / Progressive High-grade Glioma Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NTL-LEES-2018-02
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: High-grade Gliomas
MeSH Terms: interventions — 14-methyl-20-oxa-5,7,14,26-tetraazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8(27),9,11,16,21,23-decaene; Administration, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 150 mg, BIW in every 28d (Experimental): TG02 capsules were given orally at 150 mg on the 1st, 4th, 8th, 11th, 15th, 18th, 22nd and 25th day, every 28 days.
  Interventions: Drug: TG02 capsules oral administration, BIW in every 28d
- 200 mg, BIW in every 28d (Experimental): TG02 capsules were given orally at 200 mg on the 1st, 4th, 8th, 11th, 15th, 18th, 22nd and 25th day, every 28 days.
  Interventions: Drug: TG02 capsules oral administration, BIW in every 28d
- 250 mg, BIW in every 28d (Experimental): TG02 capsules were given orally at 250 mg on the 1st, 4th, 8th, 11th, 15th, 18th, 22nd and 25th day, every 28 days.
  Interventions: Drug: TG02 capsules oral administration, BIW in every 28d

INTERVENTIONS:
Drug: TG02 capsules oral administration, BIW in every 28d — TG02 capsules150mg oral administration, BIW in every 28d
  Arms: 150 mg, BIW in every 28d
Drug: TG02 capsules oral administration, BIW in every 28d — TG02 capsules 200mg oral administration, BIW in every 28d
  Arms: 200 mg, BIW in every 28d
Drug: TG02 capsules oral administration, BIW in every 28d — TG02 capsules 250mg oral administration, BIW in every 28d
  Arms: 250 mg, BIW in every 28d

SUMMARY:
The aim of the study was to explore the dose-limiting toxicity (DLT) and the maximum tolerable dose (MTD) of oral administration of TG02 capsules twice a week for 4 weeks.

DETAILED DESCRIPTION:
Using the traditional 3 +3 design, 150 mg as the initial dose and 50 mg as the increasing interval of up to 250 mg, and oral administration on the 1st, 4th, 8th, 11th, 15th, 18th, 22nd and 25th day of each 28-day cycle. Phase I clinical study to evaluate the tolerance and pharmacokinetic parameters of oral TG02 capsules.

ELIGIBILITY:
Inclusion criteria:

1. Age: 18 ~ 75 years old, both men and women.
2. Histologically proven glioblastoma or anaplastic astrocytoma that has failed from temozolomide treatment in the past.
3. According to RANO criteria, patients with clinically evaluated recurrence or progression with clearly measurable lesions.
4. If previous radiotherapy has been performed, it must be completed for a period of more than 3 months, or within 3 months but tumor progression occurs in the original radiation field or has been confirmed by histopathology. .
5. The first day of treatment was ≥ 2 weeks from the second surgery of recurrence, and the incision is healed in grade A.
6. ECOG 0 - 2 points, can swallow the drug and maintain oral administration.
7. The expected survival time was more than 3 months.
8. The hematopoietic function of bone marrow was adequate: ANC≥1.5×109/L，PLT≥100×109/L，Hb≥90 g/L；.
9. Patients who had previously undergone surgical resection were able to provide no less than 15 tumor tissue sections and pathological reports for the study.

Exclusion criteria

1. Other cytotoxic drugs were received within 28 days prior to the start of the study, or adverse reactions from previous systematic treatment have not recovered (except alopecia and pigmentation).
2. Bevacizumab was treated within 6 weeks before the start of the study.
3. Previous treatment with carmostine sustained-release implants or intracerebral implantation of radiotherapy.
4. A patient with a major seizure that cannot be effectively controlled by drugs.
5. MRI examinations cannot be performed (e.g. pacemakers, undesirable metal dentures, etc.).
6. Patients with severe impairment of liver and kidney function: ALT ≥ 2.5 ULN,AST ≥ 2.5 ULN in patients without liver metastasis; ALT ≥ 5 ULN,AST ≥ 5 ULN in patients with liver metastasis; Or TBIL ≥ 1.5 ULN, or Cr ≥ 1.5 ULN, or creatinine clearance ≤ 60 ml/ min calculated by Cockcroft-Gault formula;
7. Unstable or uncontrollable diseases or conditions related to or affecting cardiac function (e.g. unstable angina pectoris, congestive heart failure [NYHA > II], uncontrolled hypertension [diastolic blood pressure > 85 mmHg; systolic blood pressure >145 mmHg]), arrhythmia or prolonged QTc interval (male > 450 Ms; female > 470ms).
8. A history of arterial thromboembolism (such as stroke, transient ischemic attack, or myocardial infarction) within 6 months. Bleeding or hypercoagulable coagulation disorder occurred within 6 months prior to the first day of the study.
9. Active peptic ulcer or inflammatory bowel disease.
10. Active hepatitis, or HIV, Treponema pallidum infection.
11. Pregnant or breastfeeding.
12. Subjects who were unable to use adequate contraception during the study and for six months after the end of the study were unable to use adequate contraception.
13. Currently participating in another clinical trial or within 30 days of the last administration of the trial drug.
14. The subjects had conditions that affected their provision of written informed consent and / or compliance with the research process.
15. There were cases in which any other investigator did not consider it appropriate to join the group.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-03-22 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 28 days after first dose
  Adverse events of level 3 or above related to the study drug occurring within 28 days after the first dose as assessed by CTCAE v5.0.
Maximal tolerable dose(MTD) | 28 days after first dose
  DLT occurs in less than 1/6 subjects, this lower dose is defined as MTD.

SECONDARY OUTCOMES:
Overall response rate（ORR） | 12 months
  proportion of patients whose best overall response during their participation in the study is either CR or PR. The best overall response is the best response recorded from first dose until disease progression.

OTHER OUTCOMES:
c-myc expression in tumor tissue | 12 months
  the relationship between c-myc expression in tumor tissue with the tumor response

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China